CLINICAL TRIAL: NCT03599154
Title: Evaluation of GEMCITEST in Patients With Pancreatic Cancer and Treated by Chemotherapy
Acronym: GEMCIPANC
Status: Completed | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: GEMCIPANC
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
Keywords: Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cancer has a 5-year overall survival rate around 5%. It is the 6th most common cancer in France (11 600 new annual cases in 2012) and the 4th leading cause of cancer deaths in France and Europe.

Many translational research has tried to identify biomarkers in pancreatic cancer. Only the expression of hENT1 evaluated on the tumor tissue with the mouse antibody seems really relevant by providing a predictive value of the effectiveness of gemcitabine adjuvant. In a metastatic situation, there is no predictive marker of the effectiveness of chemotherapy treatments.

GemciTest(TM), studied in this study, is developed by the company Acobiom. Test based on the qRT-PCR technology that allows the establishment of a molecular signature of 10 genes that showed its interest as a biomarker in 60 patients with metastatic pancreatic adenocarcinoma treated with gemcitabine. Retrospective analysis differentiated 2 patient populations:

* 22 patients with a "favorable" expression gene with a median survival of 14.9 months
* 35 patients with an "adverse" expression gene with a median survival of 5.1 months

Primary objective: To evaluate in patients with pancreatic cancer, treated with Gemcitabine alone or combined (nab-paclitaxel) or with Folfirinox, the prognostic value of the GemciTest(TM) test on overall survival and response to treatment.

To realize this study, only one 2.5 mL blood sample is taken before starting chemotherapy. The standard practice data is then saved.

100 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed pancreatic cancer
2. Patient seeking first-line chemotherapy for pancreatic cancer
3. Age> 18 years
4. Presence of at least 1 measurable tumor lesion according to RECIST 1.1 criteria
5. Performance index ≤ 2
6. Patient able and willing to comply with the study procedures according to the protocol
7. Patient able to understand, sign and date informed consent
8. Affiliation to a social security scheme.

Exclusion Criteria:

1. Contraindication to chemotherapy
2. Anti-tumor therapy, experimental or not, recent in the last 4 weeks before the inclusion of the patient
3. Active infection requiring antibiotics within 14 days before inclusion
4. Patients unable to understand, read and / or sign informed consent
5. Persons benefiting from a protection system for adults (including tutorship and guardianship)
6. Pregnant or lactating women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with pancreatic cancer
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Overall survival | average of 1 year
  Overall survival is defined as survival between Day 1 of the first line of chemotherapy and death

CONTACTS AND LOCATIONS:
Overall Officials: François Ghiringhelli, PU PH, Study Director — Centre Georges François Leclerc, DIJON
Locations (1):
- Centre Georges François Leclerc, Dijon, France